CLINICAL TRIAL: NCT00718315
Title: A Randomized, Open Label Study to Compare the Use of the Dermatological Creams Verutex, Eritex and Fisiogel in the Management of Skin Rash Associated With Tarceva Treatment in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer.
Brief Title: A Study of Verutex (Fusidic Acid), Eritex (Erythromycin) and Fisiogel in the Management of Tarceva-Associated Rash.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21450
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Fusidic Acid; Erythromycin

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: erlotinib [Tarceva]; Drug: fusidic acid [Verutex]
- 2 (Experimental)
  Interventions: Drug: erlotinib [Tarceva]; Drug: erythromycin [Eritex]
- 3 (Experimental)
  Interventions: Drug: erlotinib [Tarceva]; Drug: Fisiogel

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150mg po daily
Drug: fusidic acid [Verutex] — topical, daily for 30 days.
  Arms: 1
Drug: erythromycin [Eritex] — topical, daily for 30 days.
  Arms: 2
Drug: Fisiogel — topical, daily for 30 days
  Arms: 3

SUMMARY:
This 3 arm study will compare the efficacy and safety of three different dermatological creams designed for prophylaxis of skin rash associated with Tarceva treatment in patients with locally advanced or metastatic non-small cell lung cancer. Eligible patients who have recently started Tarceva treatment will be randomized to one of 3 groups, to receive daily treatment with Verutex, Eritex or Fisiogel cream for 30 days, and the incidence and severity of skin rash will be assessed. The anticipated time on study treatment is <3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* locally advanced or metastatic non-small cell lung cancer (stage IIIB/IV);
* eligible to start treatment with Tarceva, or receiving Tarceva for <=5 days.

Exclusion Criteria:

* presence of skin rash or other signs of skin toxicity;
* treatment with any systemic or intranasal antibiotic within 7 days before randomization;
* treatment with other topical formulation within 14 days before randomization;
* other anticancer therapy in addition to Tarceva.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- Brazil (15):
  - Fortaleza, Ceará
  - Salvador, Estado de Bahia
  - Taguatinga, Federal District
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Divinópolis, Minas Gerais
  - Curitiba, Paraná
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Natal, Rio Grande do Norte
  - Ijuí, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Itajaí, Santa Catarina
  - Ribeirão Preto, São Paulo
  - São Paulo, São Paulo

RESULTS

PARTICIPANT FLOW:
Groups:
- Fisiogel: Participants received erlotinib 150 milligrams (mg) daily and A thin film of the topical formulation of Fisiogel was applied to face, neck, and anterior and posterior chest twice daily (every 12 hours), as per medical guidance daily for 30 days.
- Stiemicyn: Participants received erlotinib 150 mg daily and a thin film of the topical formulation of Stiemicyn was applied to face, neck, and anterior and posterior chest twice daily (every 12 hours), as per medical guidance daily for 30 days.
- Verutex: Participants received erlotinib 150 mg daily and a thin film of the topical formulation of Verutex was applied to face, neck, and anterior and posterior chest twice daily (every 12 hours), as per medical guidance daily for 30 days.
Period: Overall Study
Arm/Group | Fisiogel | Stiemicyn | Verutex
Started | 67 | 67 | 67
Completed | 48 | 45 | 46
Not Completed | 19 | 22 | 21
Not completed — Adverse Event | 1 | 2 | 3
Not completed — Death | 6 | 6 | 5
Not completed — Lost to Follow-up | 2 | 3 | 4
Not completed — Protocol Violation | 5 | 5 | 3
Not completed — Erlotinib dose decreased | 4 | 3 | 1
Not completed — Use of Minocyclin | 1 | 1 | 1
Not completed — Disease progression | 0 | 1 | 1
Not completed — Other | 0 | 0 | 1
Not completed — Use of ATB and Corticoids | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) population covered all participants who had at least one application of study drug and who had at least one post-treatment assessment, irrespective of compliance extent with protocol criteria.
Groups:
- Fisiogel: Participants received erlotinib 150 mg daily and A thin film of the topical formulation of Fisiogel was applied to face, neck, and anterior and posterior chest twice daily (every 12 hours), as per medical guidance daily for 30 days.
- Total: Total of all reporting groups
Arm/Group | Fisiogel | Stiemicyn | Verutex | Total
Number analyzed (Participants) | 67 | 67 | 67 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (11.1) | 63.6 (11.0) | 64.6 (14.0) | 64.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 31 | 26 | 94
  Male | 30 | 36 | 41 | 107

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Develop Skin Rash
Description: Skin rash was assessed by the investigator and dermatologists (the latter ones only through pictures) and scored according to (National cancer Institute -Common Terminology Criteria for Adverse Events ) NCI-CTCAE ( version 3 (line "Rash/desquamation" - short name "rash").
Time Frame: 30 Days
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fisiogel | Stiemicyn | Verutex
Number analyzed (Participants) | 65 | 65 | 67
percentage of participants | 60.0 [47.1 to 72.0] | 69.2 [56.6 to 80.1] | 73.1 [60.9 to 83.2]
Statistical Analysis 1: Comparison: Fisiogel; Test type: Superiority or Other; p = 0.481, t-test, 1 sided — Test for Binomial Ratio, where H0: P >=61%; Ha: P < 61% (One-tailed Test)
Statistical Analysis 2: Comparison: Stiemicyn; Test type: Superiority or Other; p = 0.933, t-test, 1 sided — Test for Binomial Ratio, where H0: P >=61%; Ha: P < 61% (One-tailed Test)
Statistical Analysis 3: Comparison: Verutex; Test type: Superiority or Other; p = 0.986, t-test, 1 sided — Test for Binomial Ratio, where H0: P >=61%; Ha: P < 61% (One-tailed Test)

2. Primary Outcome: Percentage of Participants With Skin Rash Stratified by Severity Grade
Description: The severity of skin rash was graded on a 5 point scale where 0 (equals)= absent, 1= mile, 2=moderate, 3= severe, 4= life threatening and 5= Death
Time Frame: 30 Days
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Fisiogel | Stiemicyn | Verutex
Number analyzed (Participants) | 57 | 60 | 60
percentage of participants
  Grade 0 | 29.8 | 25.0 | 18.3
  Grade 1 | 21.1 | 18.3 | 43.3
  Grade 2 | 49.1 | 56.7 | 35.0
  Grade 3 | 0 | 0 | 3.3
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

3. Secondary Outcome: Time to Appearance of Skin Rash
Description: Time to occurence of skin rash was calculated as the number of days from Day 0 until the first appearance of skin rash as defined by NCI-CTCAE
Time Frame: Days 0, 15, and 30
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fisiogel | Stiemicyn | Verutex
Number analyzed (Participants) | 65 | 65 | 67
Days | 16.0 [15.0 to 28.0] | 15.0 [15.0 to 16.0] | 15.0 [14.0 to 15.0]
Statistical Analysis 1: Comparison: Fisiogel vs Stiemicyn vs Verutex; Test type: Superiority or Other; p = 0.095, Log Rank

4. Secondary Outcome: Percentage of Participants With Erythema
Description: Erythema is defined as redness of the skin or mucous membranes, caused by hyperemia of superficial capillaries
Time Frame: Days 0, 15, and 30
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fisiogel | Stiemicyn | Verutex
Number analyzed (Participants) | 67 | 67 | 67
percentage of participants | 56.7 [44.8 to 67.9] | 56.7 [44.8 to 67.9] | 43.3 [32.1 to 55.2]
Statistical Analysis 1: Comparison: Fisiogel vs Stiemicyn vs Verutex; Test type: Superiority or Other; p = 0.199, Chi-squared

5. Secondary Outcome: Percentage of Participants With Pruritus
Description: Pruritus is defined as intense localized itching
Time Frame: Days 0, 15, and 30
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fisiogel | Stiemicyn | Verutex
Number analyzed (Participants) | 61 | 63 | 61
percentage of participants | 36.1 [25.2 to 48.6] | 47.6 [35.8 to 59.7] | 29.5 [19.6 to 41.9]
Statistical Analysis 1: Comparison: Fisiogel vs Stiemicyn vs Verutex; Test type: Superiority or Other; p = 0.108, Chi-squared

6. Secondary Outcome: Percentage of Participants With Pain
Description: Pain is defined as an unpleasant feeling often caused by intense or damaging stimuli
Time Frame: Days 0, 15, and 30
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fisiogel | Stiemicyn | Verutex
Number analyzed (Participants) | 67 | 67 | 67
percentage of participants | 16.4 [9.4 to 27.1] | 25.4 [16.5 to 36.9] | 13.4 [7.2 to 23.6]
Statistical Analysis 1: Comparison: Fisiogel vs Stiemicyn vs Verutex; Test type: Superiority or Other; p = 0.179, Chi-squared

7. Secondary Outcome: Percentage of Participants With Erythema Stratified by Severity Grade
Description: The severity of skin rash was graded on a 5 point scale where 0 (equals)= absent, 1= mile, 2=moderate, 3= severe, 4= life threatening and 5= Death; Severity graded by oncologist.
Time Frame: 30 Days
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Fisiogel | Stiemicyn | Verutex
Number analyzed (Participants) | 61 | 63 | 61
percentage of participants
  Grade 0 | 37.7 | 39.7 | 52.5
  Grade 1 | 39.3 | 36.5 | 39.3
  Grade 2 | 23.0 | 22.2 | 6.6
  Grade 3 | 0 | 1.6 | 1.6
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Fisiogel vs Stiemicyn vs Verutex; Test type: Superiority or Other; p = 0.066, Kruskal-Wallis

8. Secondary Outcome: Percentage of Participants With Pruritus Stratified by Severity Grade
Description: as for outcome 7
Time Frame: 30 Days
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Fisiogel | Stiemicyn | Verutex
Number analyzed (Participants) | 61 | 63 | 61
percentage of participants
  Grade 0 | 63.9 | 52.4 | 70.5
  Grade 1 | 19.7 | 31.7 | 24.6
  Grade 2 | 14.8 | 14.3 | 3.3
  Grade 3 | 1.6 | 1.6 | 1.6
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Fisiogel vs Stiemicyn vs Verutex; Test type: Superiority or Other; p = 0.087, Kruskal-Wallis

9. Secondary Outcome: Percentage of Participants With Pain Stratified by Severity Grade
Description: The severity of pain was graded on a 5 point scale where 0 (equals)= absent, 1= mile, 2=moderate, 3= severe, 4= life threatening and 5= Death; Severity graded by oncologist.
Time Frame: 30 Days
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Fisiogel | Stiemicyn | Verutex
Number analyzed (Participants) | 61 | 63 | 61
percentage of participants
  Grade 0 | 82.0 | 73.0 | 85.2
  Grade 1 | 11.5 | 22.2 | 6.6
  Grade 2 | 4.9 | 4.8 | 6.6
  Grade 3 | 1.6 | 0 | 1.6
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Fisiogel vs Stiemicyn vs Verutex; Test type: Superiority or Other; p = 0.308, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from Day 0 to Day 45 (15 days after the End of study)
Arm/Group | Fisiogel | Stiemicyn | Verutex
Serious Adverse Events (participants affected / at risk) | 12/67 | 13/66 | 19/67
Other Adverse Events (participants affected / at risk) | 45/67 | 45/66 | 48/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fisiogel (N=67) | Stiemicyn (N=66) | Verutex (N=67)
Fatigue (asthenia, lethargy, malaise (General disorders) | 0 | 2 | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 | 0 | 0
Fever (in the absence of neutropenia, where neurtropenia is defined as ANC <1.0x109/L) (General disorders) | 0 | 0 | 1
No specification (General disorders) | 0 | 1 | 0
Death not associated with CTCAE term (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2
Death not associated with CTCAE term - "cardiac arrest" (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ascites (non-malignant) (Gastrointestinal disorders) | 0 | 0 | 1
Obstruction, GI - small bowel NOS (Gastrointestinal disorders) | 1 | 0 | 0
No specification (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhage, pulmonary/upper respiratory, bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hemorrhage, GI, lower GI NOS (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage, GI, stomach (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhage, pulmonary/upper respiratory, respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Lung (pneumonia) (Infections and infestations) | 1 | 1 | 1
Pulmonary/upper respiratory (Infections and infestations) | 0 | 0 | 3
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 0 | 0
Confusion (Nervous system disorders) | 0 | 0 | 1
No specification, pulmonary/upper respiratory, pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
No specification, cardiovascular, pain (Vascular disorders) | 0 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
No specification (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 0 | 1
Vessel injury - vein - SVC (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fisiogel (N=67) | Stiemicyn (N=66) | Verutex (N=67)
Diarrhea (Gastrointestinal disorders) | 15 | 18 | 14
Anorexia (Gastrointestinal disorders) | 5 | 7 | 6
Nausea (Gastrointestinal disorders) | 3 | 4 | 3
Mucositis/stomatitis (clinical exam) - oral cavity (Gastrointestinal disorders) | 2 | 5 | 2
Vomiting (Gastrointestinal disorders) | 2 | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 2
Mucositis/stomatitis (functional/symptomatic) - oral cavity (Gastrointestinal disorders) | 2 | 1 | 1
No specification (Gastrointestinal disorders) | 0 | 1 | 3
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 | 2 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 0
No specification (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 | 8 | 4
Fever (General disorders) | 2 | 1 | 2
No specification (Skin and subcutaneous tissue disorders) | 2 | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Nail change (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Lung (pneumonia) (Infections and infestations) | 1 | 1 | 1
Pulmonary/upper respiratory (Infections and infestations) | 1 | 4 | 6
Renal/genitourinary (Infections and infestations) | 1 | 0 | 3
No specification (Infections and infestations) | 1 | 1 | 2
No specification (Gastrointestinal disorders) | 2 | 1 | 1
No specification (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
No specification (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
No specification (General disorders) | 3 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 2
Death not associated with CTCAE term (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2
Dry eye syndrome (Eye disorders) | 2 | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 2 | 2
No specification (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.